CLINICAL TRIAL: NCT00013728
Title: Asthma & Exposure to Peaks in Particulate Air Pollution
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 6214-CP-001
Record Dates: First submitted 2001-03-28; First posted 2001-03-30 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2006-03

CONDITIONS: Asthma
Keywords: asthma; particulate matter
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
We are testing the following two hypotheses: 1) Peaks in hourly exposures to airborne particulate matter (PM) of outdoor origin will be more closely associated with acute asthmatic responses to particles than 24-hour average exposures in susceptible individuals; 2) Personal exposure to PM, and estimated particle dose to the lungs, will be more closely associated with daily asthma severity than standard outdoor particle concentrations measured as 24-hour averages at governmental monitoring sites.

DETAILED DESCRIPTION:
We are testing the following two hypotheses: 1) Peaks in hourly exposures to airborne particulate matter (PM) of outdoor origin will be more closely associated with acute asthmatic responses to particles than 24-hour average exposures in susceptible individuals; 2) Personal exposure to PM, and estimated particle dose to the lungs, will be more closely associated with daily asthma severity than standard outdoor particle concentrations measured as 24-hour averages at governmental monitoring sites. Toxicological data for asthma exacerbations from particulate matter (PM) suggests that particle deposition in the lower respiratory tract can cause inflammatory and lung function changes suggestive of asthma pathology. There is now a scientific need to explain epidemiological findings of ambient PM effects on asthmatics at mass concentrations below what is expected (from toxicological data) to be harmful. One possibility is that study participants are encountering unmeasured short-term excursions of particle mass levels capable of inducing adverse reactions in the lung, but this effect is only captured somewhat by the regulatory standard of 24-hour averages. Our research in southern California is vital to the current controversy regarding regulatory standards given that a health-based scientific rationale for any specific PM averaging time is not established.

ELIGIBILITY:
1) physician-diagnosed asthma, at least a 1 yr. history, including episodic symptoms of wheezing, cough and dyspnea; 2) mild to moderate severity of asthma: i) a history of at least several weeks during the warm seasons (Mar-Oct) during which the subject required regular daily use of prescribed prophylactic asthma medications; & ii) asthma exacerbations at least 2 days/week requiring as-needed bronchodilators during an extended period of 1-2 warm season months; 3) age from 9-18; 4) home, school or work addresses in Alpine, CA area; 5) no history of smoking by the subjects and no person smoking in the subject?s home.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24
Dates: Start 2000-09; Study Completion 2003-10